CLINICAL TRIAL: NCT00716196
Title: A Prospective Study of Thin Prep Versus Papanicolau in Suspected Malignant Lesions During EUS
Brief Title: A Prospective Study of Thin Prep Versus Papanicolau in Suspected Malignant Lesions During Endoscopic Ultrasound (EUS)
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Dr. Julia LeBlanc, MD, MPH, Indiana University, Department of Medicine
Other Study IDs: 0502-23
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Suspected Malignant Lesions
Keywords: thin prep; EUS

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: The purpose of this study was to compare the performance of the monolayer preparation (Cyto Lyt or Thin prep) to the routine use of Papanicolau methods on the analysis of specimens obtained using EUS-FNA.

DETAILED DESCRIPTION:
Introduction: The presence of a pathologist during an endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) is often a luxury. In addition, preparation of multiple slides for a fine needle aspiration can be time-consuming for the gastroenterologist who waits for verbal feedback on the adequacy of the specimen. Often, a timely diagnosis is needed to direct patient management. Currently, there is no established standard of care for EUS-FNA preparation. A liquid based cytologic fixative preparation (Thin-prep or CytoLyt), is a well-established process used by pathologists for evaluating cervical smears. It has not yet been adopted or accepted for EUS-FNA. This method combines multiple aspirates on a single slide, thereby decreasing the number of slides that need to be processed and interpreted by the pathologist

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known or suspected malignancy (solid mass or lymph node) that are undergoing EUS will be eligible to participate in this study.
* Target lesions such as ascites and cystic lesions will not be considered for this study. However, if a patient has an abnormal solid lesion and abnormal lymph node in addition to the ascites or cystic lesion, they may still be considered for the study. That is, the solid lesions and abnormal lymph nodes are appropriate target lesions for this study.
* No evidence of dementia or altered mental status that would prohibit the giving and understanding of informed consent, and no evidence of psychiatric risk that would preclude adequate compliance with this protocol.
* Subject must provide signed written informed consent.

Exclusion Criteria:

* Subjects that have had a previous EUS-FNA are eligible for this study
* Target lesions such as ascites and cystic lesions will not be considered for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sample from patients presenting at the GI endoscopy unit for an EUS.
Sampling Method: Non-Probability Sample
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia K LeBlanc, MD, MPH, Principal Investigator — Indiana University
Locations (1):
- Clarian/Indiana University Hospital, Indianapolis, Indiana, United States